CLINICAL TRIAL: NCT03600376
Title: Phase 3, Multi-Center, Double-Blind, Randomized, 2-Arm, Parallel Study to Assess the Efficacy and Safety of Ryanodex (EGL-4104) as Adjuvant Treatment in Subjects With Exertional Heat Stroke (EHS)
Brief Title: Study to Assess the Efficacy and Safety of Ryanodex as Adjuvant Treatment in Subjects With EHS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eagle Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EGL-4104-C-1801
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Exertional Heat Stroke
MeSH Terms: interventions — Dantrolene; Standard of Care

STUDY DESIGN:
Intervention Model Description: Ryanodex (dantrolene sodium) for injectable suspension plus Standard of Care
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ryanodex and Standard of Care (Experimental): In addition to Standard of Care measures, Ryanodex (dantrolene sodium) for injectable suspension; 250 mg/vial will be administered.
  Interventions: Drug: Ryanodex and Standard of Care
- Standard of Care only (SOC) (Other): Standard of Care treatment will consist of the immediate start of cooling measures.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Ryanodex and Standard of Care — Ryanodex to be administered as a rapid IV push
  Other Names: Ryanodex and SOC
  Arms: Ryanodex and Standard of Care
Other: Standard of Care — Body cooling measures and supportive measures
  Other Names: SOC
  Arms: Standard of Care only (SOC)

SUMMARY:
A double-blind, parallel study of Ryanodex for the adjuvant treatment of exertional heat stroke (EHS) compared to current Standard of Care (SOC) for EHS.

DETAILED DESCRIPTION:
Following triage and primary assessment in the emergency medical facility, subjects will be randomized to 1 of 2 treatment arms, SOC plus Ryanodex or SOC only. Subjects will be dosed and followed for up to 6 hours post-randomization. Current SOC is limited to body cooling and supportive measures.

ELIGIBILITY:
Inclusion Criteria: Core body temperature of greater than or equal to 40.0 degrees C (104 degrees F); recent history of exertional activity; GCS score less than 13; tachycardia -

Exclusion Criteria: clinical severe infection; hyperthermia secondary to another condition; endotracheal intubation;; sedative drugs administered prior to or at time of study entry; likelihood of head trauma within 6 months pre-study; positive pregnancy test; history of myocardial infection within 30 days; history of seizure disorder or epilepsy; concomitant or prior use of calcium channel blockers.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-19 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hepner, Study Director — Eagle Pharmaceuticals, Inc.
Locations (4):
- Saudi Arabia (4):
  - King Faisal Hospital, Mecca
  - Mina al Jisr Hospital, Miná
  - Mina Al-Shari Al-Jadeed Hospital, Miná
  - Mina Al-Wadi Hospital, Miná

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fisher JD, Shah AP, Norozian F. Clinical Spectrum of Pediatric Heat Illness and Heatstroke in a North American Desert Climate. Pediatr Emerg Care. 2022 Feb 1;38(2):e891-e893. doi: 10.1097/PEC.0000000000002438. PMID 33848093

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ryanodex and Standard of Care | Standard of Care Only (SOC)
Started | 9 | 8
Completed | 7 | 2
Not Completed | 2 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Transferred to other facility | 1 | 0
Not completed — Investigator Decision | 0 | 4
Not completed — Determined to be ineligible for study | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ryanodex and Standard of Care | Standard of Care Only (SOC) | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (7.2) | 53.4 (11.2) | 54.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 0 | 3
  Unknown or Not Reported | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 9 | 8 | 17
Weight [Mean (Standard Deviation); unit: kg] | 86.1 (16.9) | 84.2 (12.9) | 85.2 (14.7)
Height [Mean (Standard Deviation); unit: cm] — Population: It was not possible to obtain accurate height measurements for several patients due to the extreme nature of their medical condition.
  cm
    number analyzed (Participants) | 8 | 6 | 14
    (all) | 162.8 (7.6) | 159.3 (7.7) | 161.3 (7.6)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: It was not possible to calculate BMI for several patients due to the extreme nature of their medical condition.
  kg/m^2
    number analyzed (Participants) | 8 | 6 | 14
    (all) | 32.4 (5.9) | 33.2 (5.7) | 32.7 (5.6)
Glasgow Coma Scale Score [Mean (Standard Deviation); unit: units on a scale] — The Glasgow Coma Scale (GCS) is a reliable and objective way of recording the initial and subsequent level of consciousness in a person after a brain injury. Higher total GCS represents a better outcome. The scores of subscales are summed to determine the total score.
  The range of total GCS score is from 3 - 15 where 13-15 is Mild; 9 - 12 is Moderate; and 3 -8 is Severe.
  units on a scale | 5.6 (2.7) | 5.5 (2.7) | 5.5 (2.6)
Rectal Temperature [Mean (Standard Deviation); unit: Degrees Celsius] | 41.8 (1.2) | 41.3 (0.9) | 41.5 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Recovery of Level of Consciousness Defined as a Glasgow Coma Scale (GCS) GCS ≥ 13 [Time Frame: 90 Minutes Post-randomization]
Description: The GCS is a validated and reliable scale to evaluate level of consciousness in patients with acute brain injury. The scale assesses 3 functions: Eye Opening, Verbal Response, and Motor Response. GCS scores range from 15 (best) to 3 (worst).
Time Frame: 90 minutes post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Ryanodex and Standard of Care | Standard of Care Only (SOC)
Number analyzed (Participants) | 9 | 8
Participants | 4 | 2

2. Secondary Outcome: Cumulative Incidence of Recovery of Level of Consciousness Defined as a Glasgow Coma Scale (GCS) Greater Than or Equal to 13 Over the Course of the Study [Time Frame: Study Duration]
Description: as for outcome 1
Time Frame: Treatment duration, up to 6 hours
Population: the outcome measure data table below is a summary of results showing the cumulative proportion of subjects achieving GCS score ≥13 post-randomization at all planned time points. Data is cumulative therefore the counts in the categories below will not add up to the Number Analyzed.
  score ≥ 13 post-randomization at all planned time points in the study is shown
Measure: Count of Participants; unit: Participants
Arm/Group | Ryanodex and Standard of Care | Standard of Care Only (SOC)
Number analyzed (Participants) | 9 | 8
Participants
  Pts. achieving GCS score ≥ 13 at 15 min post-randomization | 1 | 0
  Pts. achieving GCS score ≥ 13 at 30 min. post-randomization | 1 | 0
  Pts. achieving GCS score ≥ 13 after 45 min. post-randomization | 1 | 0
  Pts. achieving GCS score ≥ 13 after 60 min. post-randomization | 2 | 1
  Pts. achieving GCS score ≥ 13 after 75 min. post-randomization | 3 | 2
  Pts. achieving GCS score ≥ 13 after 90 min. post-randomization | 4 | 2
  Pts. achieving GCS score ≥ to 13 after 2 hr.. post-randomization | 5 | 2
  Pts. achieving GCS score ≥ 13 after 4 hr. post-randomization/follow-up phase | 5 | 2
  Pts. achieving GCS score ≥ 13 at end of study or early termination | 5 | 2

ADVERSE EVENTS:
Time Frame: Adverse events data was collected from time of randomization through end of study (6 hours post-randomization) or early termination.
Arm/Group | Ryanodex and Standard of Care | Standard of Care Only (SOC)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/8
Other Adverse Events (participants affected / at risk) | 7/9 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ryanodex and Standard of Care (N=9) | Standard of Care Only (SOC) (N=8)
Coma Scale Abnormal (Investigations) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ryanodex and Standard of Care (N=9) | Standard of Care Only (SOC) (N=8)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coma Scale Abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 3 (3)
Agitation (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs are not permitted to discuss or publish study results.

DOCUMENTS (2):
  • Study Protocol (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT03600376/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT03600376/SAP_001.pdf